CLINICAL TRIAL: NCT03701776
Title: Effects of Aerobic Exercise Verse Balance Training on Degenerative Cerebellar Disease
Brief Title: Ataxia and Exercise Disease Using MRI and Gait Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Scott Barbuto, Assistant Professor of Physical Medicine and Rehabilitation, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS0414
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Ataxia; Spino Cerebellar Degeneration; Spinocerebellar Ataxias
Keywords: Ataxia, exercise, spinocerebellar disease, neuroimaging
MeSH Terms: conditions — Ataxia; Spinocerebellar Degenerations; Spinocerebellar Ataxias; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single blind randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will know that the participant has received balance or aerobic training, but will not be aware of which group the participant belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training (Experimental): Participants will be given a stationary exercise bike for home use. They will be instructed to use the exercise bike five times a week for thirty-minute sessions. The exercise intensity prescription will be based on the subject's VO2max determined on pre-test day. The exercise program will start at 60% of intensity per session, and then will be increased by steps of 5% intensity every 2 sessions until participants reach 30 minutes of training at 80% intensity. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be instructed to log each training session. Subjects will record duration of exercise, perceived exertion, average heart rate, maximum heart rate, and distance.
  Interventions: Behavioral: Aerobic Training
- Balance Training (Active Comparator): A physical therapist will tailor a home balance training program for each participant based on pre-training capabilities. Subjects will be asked to perform exercises five times a week for thirty-minute sessions. Both dynamic and static exercises will be performed in sitting and standing positions. Exercises will start with stabilizing in a challenging static position and progress to dynamic arm and leg movements in the same or modified position. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be required to log their exercise effort in terms of frequency and level of balance challenge. Individuals will be instructed to perform more difficult exercises if balance challenge scores are low.
  Interventions: Behavioral: Balance Training

INTERVENTIONS:
Behavioral: Aerobic Training — Aerobic training on stationary bicycle for 30 minutes a day, 5 days a week for 6 months
  Arms: Aerobic Training
Behavioral: Balance Training — Standard of care
  Arms: Balance Training

SUMMARY:
The first aim is to show balance training improves DCD individual's ability to compensate for their activity limitations, but does not impact disease progression.

The second aim is to demonstrate aerobic exercise improves balance and gait in DCD persons by affecting brain processes and slowing cerebellar atrophy.

DETAILED DESCRIPTION:
Individuals with degenerative cerebellar disease (DCD) exhibit gradual loss of coordination resulting in impaired balance, gait deviations, and severe, progressive disability. With no available disease-modifying medications, balance training is the primary treatment option to improve motor skills and functional performance. There is no evidence, however, that balance training impacts DCD at the tissue level.

Aerobic training, on the other hand, may modify DCD progression as evident from animal data. Compared to sedentary controls, aerobically trained DCD rats have enhanced lifespan, motor function, and cerebellar Purkinje cell survival. Numerous animal studies also document that aerobic training has a direct, favorable effect on the brain that includes production of neurotrophic hormones, enhancement of neuroplasticity mechanisms, and protection from neurotoxins.

The effects of aerobic training in humans with DCD are relatively unknown, despite these encouraging animal data. A single study to date has evaluated the benefits of aerobic exercise on DCD in humans, and this was a secondary outcome of the study. Although participants performed limited aerobic training during the study, modest functional benefits were still detected.

The main objective of this project will be to compare the benefits of aerobic versus balance training in DCD. We hypothesize that both aerobic and balance training will improve function in DCD subjects, but that the mechanisms in which these improvements occur differ. 1) Balance training improves DCD individual's ability to compensate for their activity limitations, but does not impact disease progression. 2) Aerobic exercise improves balance and gait in DCD persons by affecting brain processes and slowing cerebellar atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spinocerebellar ataxia
* Cerebellar atrophy on MRI
* Prevalence of ataxia on clinical exam
* Ability to safely ride a stationary exercise bike

Exclusion Criteria:

* Other neurologic conditions
* Heart disease
* Cognitive impairment
* Medical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in SARA scores | 6 months
  Ataxia severity will be measured using the Scale for the Assessment and Rating of Ataxia (SARA).17 SARA evaluates the degree of ataxia by measuring gait, stance, sitting balance, speech, finger-chase test, nose-finger test, fast alternating movements, and heel-shin test.

SECONDARY OUTCOMES:
Change in gait parameters | 6 months
  For the walking assessment, participants will walk as fast as possible on a 10-meter runway six times, and we will average the times of trials 3-6. We will also collect marker position data from infrared emitting diodes placed bilaterally at the first and fifth metatarsal heads, heels, medial and lateral malleoli, medial and lateral condyles of the knee, head of the fibula, and anterior and posterior superior iliac crests pelvic crests using a three-dimensional Vicon motion capture system (Vicon, Denver, CO). Custom Nexus and Bodybuilder software will be used to calculate joint position and determine the following walking parameters: stride length, stride length variability, percent time in double limb support, and degree of pelvic rotation and tilt.
Change in cerebellar volume | 6 months
  Cranial MRI will be performed in all participants using a 3-T scanner. Using each individual's T1-weighted image, structural imaging measures of cerebellar brain volume will be derived using the FreeSurfer software package (http://surfer.nmr.mgh.harvard.edu/). FreeSurfer will automatically assign a neuroanatomic label to each voxel. From this labeling, a set of volumetric regions of interest is defined. The calculated volume within the cerebellar region is adjusted for variations in individual's intracranial brain volume (ICV) which is measured using BrainWash (an automatic multi-atlas skull-striping software package). We will process the longitudinal T1-weighted images using FreeSurfer longitudinal pipeline, recently implemented to detect small or subtle changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Barbuto, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University/New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbuto S, Kuo SH, Winterbottom L, Lee S, Stern Y, O'Dell M, Stein J. Home Aerobic Training for Cerebellar Degenerative Diseases: a Randomized Controlled Trial. Cerebellum. 2023 Apr;22(2):272-281. doi: 10.1007/s12311-022-01394-4. Epub 2022 Mar 18. PMID 35303255